CLINICAL TRIAL: NCT05552768
Title: Effects of Supracrestal Tissue Attachment Dimensions on Peri-implant Health: A RCT
Brief Title: Supracrestal Tissue Attachment Dimensions & Peri-implant Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MIS Implant Technologies, Ltd (Industry)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIS2021-01
Record Dates: First submitted 2022-09-15; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Dental Implant Placement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bone level-driven placement (BL Group) (Active Comparator): Implants will be placed at the bone level, they will receive a 1.5-2 mm long CONNECT abutment.
  Interventions: Procedure: Bone level-driven placement
- Biological width-driven placement guidelines (BW Group) (Experimental): Implants will be placed 4 mm below the mucosal margin using a 2-3 mm long CONNECT abutment.
  Interventions: Procedure: Biological width-driven placement guidelines

INTERVENTIONS:
Procedure: Bone level-driven placement — The objective of this study will be to determine if implants placed according to the soft tissue-driving implant placement paradigm, i.e. 4 mm below the tissue margin will have different clinical performance as compared to the bone level-driven placement paradigm.
  Arms: Bone level-driven placement (BL Group)
Procedure: Biological width-driven placement guidelines — Biological width-driven placement guidelines
  Arms: Biological width-driven placement guidelines (BW Group)

SUMMARY:
Decision making in regards to the 3D implant positioning in partially edentulous sites is a complex process particularly when there are adjacent teeth present. Presently, the prevailing paradigm of implant placement guidelines is bone-driven. It calls to seat the implant neck in a crestal position. Clinical studies have demonstrated that implants placed in sites with thin soft tissues are suffering more crestal bone loss than sites with thick gingiva. Consequently, it has been proposed either to place these implants in a subcrestal position or to thicken locally the soft tissues. A recommendation of how much subcrestally the implants should be inserted in these sites is still lacking but clinicians empirically implement a deeper insertion of 1.5-2 mm under the crest. There is some indication that subcrestal placement may lead to bone remodeling above the implant neck and limited bone loss beyond the neck, but clinical trials of bone level implants have not been performed to answer this definitively.

Evolving data on the dimensions of the supracrestal tissue attachment zone (aka biological width, BW) around implants suggest that a distance of 4 mm is reserved to accommodate for junctional epithelial and connective tissue attachment zones as well as a healthy peri-implant sulcus. The objective of this study will be to determine if implants placed according to the soft tissue-driving implant placement paradigm, i.e. 4 mm below the tissue margin and associated with a deeper mucosal tunnel will have less bone loss but a more compromised peri-implant health as compared to implants placed at the bone crest level following the bone-driven implant placement paradigm with more bone loss but a shallower mucosal tunnel.It is hypothesized that using the CONNECT as a dedicated immediate tissue-level abutment system which enables avoiding alteration of the peri-implant gingival seal, both groups, the one with a deeper mucosal tunnel and the one with a shallower one, will perform identical in terms of peri-implant health and tissue maintenance outcomes. This would then justify the safe placement of implants in a biologically appropriate manner using biological width-driven placement guidelines.

To test this hypothesis, two groups of 30 patients each will be treated according to either the bone-driven or the soft tissue-driven concepts:

Control group following the bone level-driven placement guidelines (BL Group): Implants will be placed at the bone level, they will receive a 1.5-2 mm long CONNECT abutment.

Test group following the biological width-driven placement guidelines (BW Group): Implants will be placed 4 mm below the mucosal margin using a 3 mm long CONNECT abutment: this means that the implant will be placed sub-crestally in agreement with the corresponding guideline, i.e. at deepest 1 mm subcrestally.

ELIGIBILITY:
Inclusion Criteria:

1. adults 21-75-year old;
2. ASA 1-3 with no medical contraindication for implant surgery;
3. Edentulous site(s) in need of implant-supported fixed restoration of one or up to three units supported by 2 implants;
4. availability of native bone of at least 6 mm in width to accommodate standard Ø 3.75 and 4.2 mm implant without any need for bone augmentation;
5. bone height to accommodate 10 mm long implants accounting for up to 2 mm of subcrestal placement in the mandible and the maxilla;
6. adequate oral hygiene and stable periodontal status with bleeding on probing (BOP) < 20% and plaque index (PI) < 30%;
7. keratinized gingiva ≥ 4 mm;
8. willing to sign an informed consent and ability and willingness to comply with all study visits.

Exclusion Criteria:

1. moderate or heavy smoking (≥10 cigarettes per day);
2. systemic diseases preventing implant placement;
3. uncontrolled diabetes (HbA1c ≥ 8%), osteoporosis as confirmed by z/t score, or other conditions or medications affecting bone healing;
4. poor oral hygiene;
5. alcoholism and recreational drug addiction;
6. uncontrolled periodontitis;
7. pregnant or lactating women;

local exclusion criteria

1. Immediate implant placement;
2. socket preservation with a bone substitute biomaterial less than 6 months prior, or 9 months prior for xenografts;
3. vertical (Seibert class II / III defect exceeding 3 mm that would compromise ideal apicocoronal placement);
4. prior ridge augmentation / GBR procedure
5. implant primary stability not enabling torquing the CONNECT abutment at 30 Ncm without rotation;

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in probing depth (PD) | 12 months post-loading

SECONDARY OUTCOMES:
Change in marginal bone levels (radiographic) | 12 months post-loading
Change in BOP | 12 months post-loading
Frequency of peri-implantitis according to the AAP classification criteria | 12 months post-loading
Number of participants with Implant Success | 12 months post-loading

CONTACTS AND LOCATIONS:
Overall Officials: Serge Szmukler, Dr, Study Director — Director of Research
Locations (1):
- Mis Implants Technologies Ltd., Misgav Regional Council, Israel

IPD SHARING:
Plan to Share IPD: Undecided